CLINICAL TRIAL: NCT05967871
Title: Pilot Feasibility Study of Fecal Microbiota Transplant for the Treatment of Small Intestinal Bacterial Overgrowth
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: McMaster Children's Hospital (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Nikhil Pai, Associate Professor, Division of Pediatric Gastroenterology & Nutrition, Hamilton Health Sciences Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16581
Record Dates: First submitted 2023-07-13; First posted 2023-08-01 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Small Intestinal Bacterial Overgrowth
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fecal Microbiota Transpant (Experimental): Participants will receive a Fecal Microbiota transplant Infusion via participants' existing enteral feeding tubes or via elective upper endoscopy (with infusion into the duodenum). Most patients with SBS at MCH and HSC have an existing enteral feeding tube (gastrostomy or jejunostomy tube).
  Interventions: Biological: Fecal Microbiota Transplant

INTERVENTIONS:
Biological: Fecal Microbiota Transplant — Participants will receive approximately 50 grams of human stool/150mL (approximately 107 microbes/mL of suspension) in saline, prepared as per standard collection, preparation, and screening protocols for FMT infusion developed by our institutional stool bank in accordance with recognized standards. Fecal microbiota transplant infused via existing enteral feeding tube or upper elective endoscopy (with infusion into the duodenum) x1.

SUMMARY:
The objective of the study is to assess feasibility, and clinical efficacy of a novel Fecal Microbiota Transplantation protocol for the treatment of pediatric small intestinal bacterial overgrowth (SIBO).

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE Fecal microbiota transplant (FMT) is an established treatment for the management of recurrent Clostridioides difficile (CDI) infection in children and adults, including children with underlying immunodeficiency syndromes and extensive surgical resection. While CDI is the most common indication for FMT, this intervention has also been studied for Crohn's disease, ulcerative colitis, autism, and small intestinal bacterial overgrowth (SIBO). SIBO is a disorder in which the small bowel is colonized by excessive aerobic and anaerobic microbes normally present in the colon. This condition may cause malabsorption, bloating, bloodstream infections (BSI), and D-lactic acidosis (DLA). Treatment traditionally involves broad-spectrum antibiotic use yet this approach may promote persistent dysbiosis, multidrug resistant organisms (MDROs), and often lacks clinical efficacy. Patients with short bowel syndrome (SBS), which involves intestinal resection, dysmotility, and altered enteral feeding are at highest risk for SIBO. Pediatric SBS SIBO patients face significant impacts on quality of life, and higher rates of bacteremia and liver disease.

Specific Aims i. To determine the feasibility, and safety of administering an FMT based treatment to pediatric SBS patients with SIBO. This aim will include measures of adverse events, acceptability to children and parents, ease of administration and sample collection.

ii. To determine short-term clinical efficacy of FMT for the treatment of SIBO. This aim will include measures of time to symptom resolution, completeness of symptom resolution, change in enteral feeding tolerance, and development of any new clinical gastrointestinal symptoms after FMT. Weeks 1-4 after FMT.

iii. To determine long-term clinical efficacy of FMT for the treatment of SIBO. This aim will include measures of durability of remission, including time to recurrence of symptom resolution, severity of clinical symptoms if recurrence, sustained changes in feeding tolerance, and efficacy of repeat FMT administration (second treatment). Week 8 after FMT.

iv. To assess changes in intestinal microbial composition and function before and after FMT. This aim will attempt to identify functional changes in the intestinal microbiome that correlate with symptom resolution. These data will support future translational and clinical studies with our collaborators and support the development of new therapeutic innovations.

D. TRIAL OBJECTIVES Our objectives are to assess feasibility, and clinical efficacy of this intervention in children (Table 2).

Feasibility Objectives:

Acceptability of this intervention for patients and families, ability of patients and families to conduct the required screening to monitor efficacy and recruitment rate of patients to the study.

Clinical Objectives:

Clinical efficacy of treating SIBO in our patient population using FMT. These outcomes will be collected at the following timepoints: baseline (pre-FMT), one-, four-, and eight-weeks post-FMT administration

E. STUDY DESIGN AND DURATION We will recruit 5-17-year-old patients with intestinal resection (any length), experiencing an active episode of SIBO (diagnosed through lactose breath testing and gastrointestinal symptom scores). Patients will discontinue antibiotics for >1 week prior to FMT. FMT infusions will be administered through patients' existing enteral tubes (gastrostomy, jejunostomy), or potentially via endoscopy (duodenal infusion).

Patients will receive a single FMT (Week 0). They will then have outcomes (including a combination of clinical symptom scores, blood, stool and urine testing) measured one week after FMT, four weeks after FMT, and eight weeks after FMT.

As this is an open-label trial, there will be no randomization or blinding required.

A placebo / comparative treatment will not be assessed.

All FMT treatments will be conducted at MCH, using local pediatric stool bank materials. Patients will have follow-up monitoring, per protocol through their local institution (MCH/HSC). Serial measurements of biological, clinical and microbial outcomes will occur, per protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients 3-18 years old
* Patients will discontinue antibiotics for at least 1 week prior to FMT
* A diagnosis of SIBO established through lactose breath test (LBT), and showing of symptoms of SIBO

Exclusion Criteria:

* Participants will not be permitted to start any new treatments (including antibiotics, probiotics, antacid treatments, or antimotility treatments) until Week 8, unless clinically indicated
* We will exclude participants <3yo to avoid potential concerns of microbial transmission in young children, and to ensure participants are developmentally able to perform LBT

  * All potential participants should request a referral through their primary, or subspecialty physician. We would be pleased to help facilitate this contact if needed, provided the appropriate contact information can be sent.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Symptoms (pre/post fecal microbiota transplant) | Baseline (pre-fecal microbiota transplant), one-, four-, and eight-weeks post-fecal microbiota transplant administration.
  SIBO Clinical Symptom Scores will be measured using the PedsQL Gastrointestinal Symptoms Scale. This validated instrument has strong age-specific test-retest properties and has been used for functional GI disorders, which have symptoms that strongly overlap with SIBO. Participants will also report symptoms using a Likert scale (Izumo scale). Results of both will be compared.
Rate of Clinical Remission (post fecal microbiota transplant) | Baseline (pre-fecal microbiota transplant), one-, four-, and eight-weeks post-fecal microbiota transplant administration.
  Absence of SIBO symptoms
Urine Metabolomics Analysis | Baseline (pre-fecal microbiota transplant), one-, four-, and eight-weeks post-fecal microbiota transplant administration.
  Collected urine will be assessed by multisegment injection-capillary electrophoresis-mass spectrometry (MSI-CE-MS), using previously described protocols. This technique will offer additional data on microbiome functional changes. Samples will be measured centrally through the Britz-McKibbin laboratory (PBM). Urine metabolomics outcomes are exploratory.
Change in Microbiome Composition, Function (pre/post fecal microbiota transplant) | Baseline (pre-fecal microbiota transplant), one-, four-, and eight-weeks post-fecal microbiota transplant administration.
  Stool will be collected for microbiome 16S rRNA and shotgun metagenomic sequencing. Samples will be obtained from either stool (per rectum), or distal ostomy outputs (ostomy in continuity with proximal bowel). All samples will be sequenced centrally through the McMaster Genomics Centre (MGC). Samples will be stored in -80 freezers. Participants unable to bring stool samples to MCH or HSC will receive funding support for temperature-controlled courier services from home. Costs of microbiome analyses will be partially subsidized by collaborators (MS).
Change in Breath Test Results (pre/post fecal microbiota transplant) | Baseline (pre-fecal microbiota transplant), one-, four-, and eight-weeks post-fecal microbiota transplant administration.
  Lactulose breath test
Bloodwork | Baseline and Week 8 (post-FMT)
  Bloodwork will include complete blood count (CBC), C-reactive protein (CRP), ferritin, folic acid, alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase (ALP), serum cytokine profiles (including IL-2, IL-6, IL10, IL-18, TNF) and serum bile acids. Routine institutional testing protocols will be followed at MCH and HSC. Bloodwork outcomes are exploratory. Data will support the development of primary and secondary objectives for future studies.

SECONDARY OUTCOMES:
Monthly Rate of Recruitment | 30 weeks
  Recruitment/month. ≥2 participants/month.
Adverse Events | 30 Weeks
  Adverse and serious events will be recorded using the Common Terminology Criteria for Adverse Events. <10% participants
Blood, stool specimens, breath tests, clinical symptom scores | 30 Weeks
  Participant provides all required blood, stool, lactulose breath tests, and symptom scores per protocol. >80% participants

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Pai, MD, Principal Investigator — McMaster Children's Hospital (McMater University)
Locations (2):
- Canada (2):
  - McMaster Children's Hospital, Hamilton, Ontario
  - Hospital for Sick Children (SickKids), Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified individual participant data (IPD) may be shared. No directly identifying information (such as names, dates of birth, contact information, or medical record numbers) will ever be disclosed. If data are shared, they will be limited to variables relevant to the outcomes reported in the trial and will be made available in de-identified form for secondary research purposes under appropriate data use agreements.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: De-identified individual participant data (IPD) and supporting documentation (such as the study protocol and statistical analysis plan) will be available beginning 12 months after publication of the primary results. Data will remain available for at least 5 years thereafter.
Access Criteria: Access will be provided to qualified researchers from academic, non-profit, or health system organizations for scientifically sound secondary analyses. Industry investigators may also request access; such requests will be considered on a case-by-case basis and granted only at the discretion of the study investigators. All data will be shared in de-identified form through a secure platform or under a data use agreement that prohibits re-identification and restricts use to the approved research purpose.

REFERENCES:
- [Background] Davidovics ZH, Michail S, Nicholson MR, Kociolek LK, Pai N, Hansen R, Schwerd T, Maspons A, Shamir R, Szajewska H, Thapar N, de Meij T, Mosca A, Vandenplas Y, Kahn SA, Kellermayer R; FMT Special Interest Group of the North American Society of Pediatric Gastroenterology Hepatology, Nutrition, the European Society for Pediatric Gastroenterology Hepatology, Nutrition. Fecal Microbiota Transplantation for Recurrent Clostridium difficile Infection and Other Conditions in Children: A Joint Position Paper From the North American Society for Pediatric Gastroenterology, Hepatology, and Nutrition and the European Society for Pediatric Gastroenterology, Hepatology, and Nutrition. J Pediatr Gastroenterol Nutr. 2019 Jan;68(1):130-143. doi: 10.1097/MPG.0000000000002205. PMID 30540704
- [Background] Nicholson MR, Mitchell PD, Alexander E, Ballal S, Bartlett M, Becker P, Davidovics Z, Docktor M, Dole M, Felix G, Gisser J, Hourigan SK, Jensen MK, Kaplan JL, Kelsen J, Kennedy M, Khanna S, Knackstedt E, Leier M, Lewis J, Lodarek A, Michail S, Oliva-Hemker M, Patton T, Queliza K, Russell GH, Singh N, Solomon A, Suskind DL, Werlin S, Kellermayer R, Kahn SA. Efficacy of Fecal Microbiota Transplantation for Clostridium difficile Infection in Children. Clin Gastroenterol Hepatol. 2020 Mar;18(3):612-619.e1. doi: 10.1016/j.cgh.2019.04.037. Epub 2019 Apr 19. PMID 31009795
- [Background] Pai N, Popov J, Hill L, Hartung E. Protocol for a double-blind, randomised, placebo-controlled pilot study for assessing the feasibility and efficacy of faecal microbiota transplant in a paediatric Crohn's disease population: PediCRaFT Trial. BMJ Open. 2019 Nov 28;9(11):e030120. doi: 10.1136/bmjopen-2019-030120. PMID 31784432
- [Background] Pai N, Popov J, Hill L, Hartung E, Grzywacz K, Moayyedi P; McMaster Pediatric Fecal Microbiota Transplant Research Collaboration. Results of the First Pilot Randomized Controlled Trial of Fecal Microbiota Transplant In Pediatric Ulcerative Colitis: Lessons, Limitations, and Future Prospects. Gastroenterology. 2021 Aug;161(2):388-393.e3. doi: 10.1053/j.gastro.2021.04.067. Epub 2021 May 4. No abstract available. PMID 33961887
- [Background] Bakker GJ, Nieuwdorp M. Fecal Microbiota Transplantation: Therapeutic Potential for a Multitude of Diseases beyond Clostridium difficile. Microbiol Spectr. 2017 Aug;5(4):10.1128/microbiolspec.bad-0008-2017. doi: 10.1128/microbiolspec.BAD-0008-2017. PMID 28840809
- [Background] Fiorentino M, Sapone A, Senger S, Camhi SS, Kadzielski SM, Buie TM, Kelly DL, Cascella N, Fasano A. Blood-brain barrier and intestinal epithelial barrier alterations in autism spectrum disorders. Mol Autism. 2016 Nov 29;7:49. doi: 10.1186/s13229-016-0110-z. eCollection 2016. PMID 27957319
- [Background] Kang DW, Adams JB, Gregory AC, Borody T, Chittick L, Fasano A, Khoruts A, Geis E, Maldonado J, McDonough-Means S, Pollard EL, Roux S, Sadowsky MJ, Lipson KS, Sullivan MB, Caporaso JG, Krajmalnik-Brown R. Microbiota Transfer Therapy alters gut ecosystem and improves gastrointestinal and autism symptoms: an open-label study. Microbiome. 2017 Jan 23;5(1):10. doi: 10.1186/s40168-016-0225-7. PMID 28122648
- [Background] Davidovics ZH, Vance K, Etienne N, Hyams JS. Fecal Transplantation Successfully Treats Recurrent D-Lactic Acidosis in a Child With Short Bowel Syndrome. JPEN J Parenter Enteral Nutr. 2017 Jul;41(5):896-897. doi: 10.1177/0148607115619931. Epub 2015 Nov 29. PMID 26616138
- [Background] Gu L, Ding C, Tian H, Yang B, Zhang X, Hua Y, Zhu Y, Gong J, Zhu W, Li J, Li N. Serial Frozen Fecal Microbiota Transplantation in the Treatment of Chronic Intestinal Pseudo-obstruction: A Preliminary Study. J Neurogastroenterol Motil. 2017 Apr 30;23(2):289-297. doi: 10.5056/jnm16074. PMID 27840368
- [Background] Bulik-Sullivan EC, Roy S, Elliott RJ, Kassam Z, Lichtman SN, Carroll IM, Gulati AS. Intestinal Microbial and Metabolic Alterations Following Successful Fecal Microbiota Transplant for D-Lactic Acidosis. J Pediatr Gastroenterol Nutr. 2018 Oct;67(4):483-487. doi: 10.1097/MPG.0000000000002043. PMID 29901551
- [Background] McGrath KH, Pitt J, Bines JE. Small intestinal bacterial overgrowth in children with intestinal failure on home parenteral nutrition. JGH Open. 2019 Apr 4;3(5):394-399. doi: 10.1002/jgh3.12174. eCollection 2019 Oct. PMID 31633044
- [Background] Thanert R, Thanert A, Ou J, Bajinting A, Burnham CD, Engelstad HJ, Tecos ME, Ndao IM, Hall-Moore C, Rouggly-Nickless C, Carl MA, Rubin DC, Davidson NO, Tarr PI, Warner BB, Dantas G, Warner BW. Antibiotic-driven intestinal dysbiosis in pediatric short bowel syndrome is associated with persistently altered microbiome functions and gut-derived bloodstream infections. Gut Microbes. 2021 Jan-Dec;13(1):1940792. doi: 10.1080/19490976.2021.1940792. PMID 34264786
- [Background] Xu F, Li N, Wang C, Xing H, Chen D, Wei Y. Clinical efficacy of fecal microbiota transplantation for patients with small intestinal bacterial overgrowth: a randomized, placebo-controlled clinic study. BMC Gastroenterol. 2021 Feb 6;21(1):54. doi: 10.1186/s12876-021-01630-x. PMID 33549047
- [Background] Allegretti JR, Kassam Z, Chan WW. Small Intestinal Bacterial Overgrowth: Should Screening Be Included in the Pre-fecal Microbiota Transplantation Evaluation? Dig Dis Sci. 2018 Jan;63(1):193-197. doi: 10.1007/s10620-017-4864-8. Epub 2017 Nov 29. PMID 29188472
- [Background] Pai N, Popov J. Protocol for a randomised, placebo-controlled pilot study for assessing feasibility and efficacy of faecal microbiota transplantation in a paediatric ulcerative colitis population: PediFETCh trial. BMJ Open. 2017 Aug 21;7(8):e016698. doi: 10.1136/bmjopen-2017-016698. PMID 28827258
- [Background] Varni JW, Bendo CB, Denham J, Shulman RJ, Self MM, Neigut DA, Nurko S, Patel AS, Franciosi JP, Saps M, Verga B, Smith A, Yeckes A, Heinz N, Langseder A, Saeed S, Zacur GM, Pohl JF. PedsQL gastrointestinal symptoms module: feasibility, reliability, and validity. J Pediatr Gastroenterol Nutr. 2014 Sep;59(3):347-55. doi: 10.1097/MPG.0000000000000414. PMID 24806837
- [Background] Maeda Y, Murakami T. Diagnosis by Microbial Culture, Breath Tests and Urinary Excretion Tests, and Treatments of Small Intestinal Bacterial Overgrowth. Antibiotics (Basel). 2023 Jan 28;12(2):263. doi: 10.3390/antibiotics12020263. PMID 36830173
- [Background] Cammarota G, Ianiro G, Tilg H, Rajilic-Stojanovic M, Kump P, Satokari R, Sokol H, Arkkila P, Pintus C, Hart A, Segal J, Aloi M, Masucci L, Molinaro A, Scaldaferri F, Gasbarrini G, Lopez-Sanroman A, Link A, de Groot P, de Vos WM, Hogenauer C, Malfertheiner P, Mattila E, Milosavljevic T, Nieuwdorp M, Sanguinetti M, Simren M, Gasbarrini A; European FMT Working Group. European consensus conference on faecal microbiota transplantation in clinical practice. Gut. 2017 Apr;66(4):569-580. doi: 10.1136/gutjnl-2016-313017. Epub 2017 Jan 13. PMID 28087657
- [Background] Food and Drug Adminstration. Guidance for Industry: Enforcement Policy Regarding Investigational New Drug Requirements for Use of Fecal Microbiota for Transplantation to Treat Clostridium Difficile Infection Not Responsive to Standard Therapies.; 2016.
- [Background] Podlesny D, Durdevic M, Paramsothy S, Kaakoush NO, Hogenauer C, Gorkiewicz G, Walter J, Fricke WF. Identification of clinical and ecological determinants of strain engraftment after fecal microbiota transplantation using metagenomics. Cell Rep Med. 2022 Aug 16;3(8):100711. doi: 10.1016/j.xcrm.2022.100711. Epub 2022 Aug 4. PMID 35931074
- [Background] Furuta K, Ishihara S, Sato S, Miyake T, Ishimura N, Koshino K, Tobita H, Moriyama I, Amano Y, Adachi K, Ohta A, Kinoshita Y. [Development and verification of the Izumo Scale, new questionnaire for quality of life assessment of patients with gastrointestinal symptoms]. Nihon Shokakibyo Gakkai Zasshi. 2009 Oct;106(10):1478-87. Japanese. PMID 19834295
- [Background] Kuehnbaum NL, Kormendi A, Britz-McKibbin P. Multisegment injection-capillary electrophoresis-mass spectrometry: a high-throughput platform for metabolomics with high data fidelity. Anal Chem. 2013 Nov 19;85(22):10664-9. doi: 10.1021/ac403171u. Epub 2013 Nov 6. PMID 24195601
- [Background] Conover KR, Absah I, Ballal S, Brumbaugh D, Cho S, Cardenas MC, Knackstedt ED, Goyal A, Jensen MK, Kaplan JL, Kellermayer R, Kociolek LK, Michail S, Oliva-Hemker M, Reed AW, Weatherly M, Kahn SA, Nicholson MR. Fecal Microbiota Transplantation for Clostridioides difficile Infection in Immunocompromised Pediatric Patients. J Pediatr Gastroenterol Nutr. 2023 Apr 1;76(4):440-446. doi: 10.1097/MPG.0000000000003714. Epub 2023 Jan 31. PMID 36720105
- [Background] Nicholson MR, Alexander E, Ballal S, Davidovics Z, Docktor M, Dole M, Gisser JM, Goyal A, Hourigan SK, Jensen MK, Kaplan JL, Kellermayer R, Kelsen JR, Kennedy MA, Khanna S, Knackstedt ED, Lentine J, Lewis JD, Michail S, Mitchell PD, Oliva-Hemker M, Patton T, Queliza K, Sidhu S, Solomon AB, Suskind DL, Weatherly M, Werlin S, de Zoeten EF, Kahn SA; North American Society of Pediatric Gastroenterology and Nutrition Faecal Microbiota Transplantation Special Interest Group. Efficacy and Outcomes of Faecal Microbiota Transplantation for Recurrent Clostridioides difficile Infection in Children with Inflammatory Bowel Disease. J Crohns Colitis. 2022 Jun 24;16(5):768-777. doi: 10.1093/ecco-jcc/jjab202. PMID 34788420
- [Background] Kunz AN, Noel JM, Fairchok MP. Two cases of Lactobacillus bacteremia during probiotic treatment of short gut syndrome. J Pediatr Gastroenterol Nutr. 2004 Apr;38(4):457-8. doi: 10.1097/00005176-200404000-00017. No abstract available. PMID 15085028
- [Background] Naranjo CA, Busto U, Sellers EM, Sandor P, Ruiz I, Roberts EA, Janecek E, Domecq C, Greenblatt DJ. A method for estimating the probability of adverse drug reactions. Clin Pharmacol Ther. 1981 Aug;30(2):239-45. doi: 10.1038/clpt.1981.154. No abstract available. PMID 7249508
- See also: US Department of Health and Human Services. Common Terminology Criteria for Adverse Events (CTCAE). Published 2017. — https://ctep.cancer.gov/protocolDevelopment/templates_applications.htm